CLINICAL TRIAL: NCT05037422
Title: Single-center Retrospective Study of the Long-term Results of the Stapled TransAnal Rectal Resection (STARR) Operation Proposed in the Treatment of a Rectocele in Consecutive Patients
Brief Title: Long-term Results of the Stapled Transanal Rectal Resection (STARR) Operation Proposed in the Treatment of a Rectocele
Acronym: STARRLOC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC21.144
Record Dates: First submitted 2021-04-29; First posted 2021-09-08 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Rectocele; Female
MeSH Terms: conditions — Rectocele

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: STARR surgery — This intervention is carried out under general anesthesia or spinal anesthesia. It consists of the circular resection of the "surplus" of rectal mucosa. Rectal resection and suturing is performed using automatic mechanical forceps introduced through the anus.

SUMMARY:
Rectal static disorders, including the rectocele, represent a frequent functional pathology which affects the quality of life of affected patients. Among vaginal treatments, the STARR technique corresponds to rectal resection by transanal approach using a stapler. The American Gastroenterology Association (AGA) has concluded that service to patients is insufficient. The technical and functional results published are mostly short-term studies. The investigators seek to assess the technical and functional results of Operation STARR, based on a series of consecutive expert center cases, to confirm or refute the conclusions of the AGA recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Patient operated for rectocele for 10 or more
* Age 18 and over
* Informed patients

Exclusion Criteria:

* Patient objection

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: All adult patients operated on for rectocele in the digestive surgery and emergency department of the CHU de Grenoble will be included, provided they are not opposed.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2021-10-16 (Actual); Primary Completion 2024-10-24 (Estimated); Study Completion 2024-11-24 (Estimated)

PRIMARY OUTCOMES:
Long term results of the STARR operation. | 10 years
  Dyschezia postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Faucheron, MD, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- CHU Grenoble Alpes, Service de chirurgie digestive et de l'urgence, Grenoble, France

REFERENCES:
- [Background] Lehur PA, Stuto A, Fantoli M, Villani RD, Queralto M, Lazorthes F, Hershman M, Carriero A, Pigot F, Meurette G, Narisetty P, Villet R; ODS II Study Group. Outcomes of stapled transanal rectal resection vs. biofeedback for the treatment of outlet obstruction associated with rectal intussusception and rectocele: a multicenter, randomized, controlled trial. Dis Colon Rectum. 2008 Nov;51(11):1611-8. doi: 10.1007/s10350-008-9378-1. Epub 2008 Jul 19. PMID 18642046
- [Background] Slim K, Mezoughi S, Launay-Savary MV, Tuech JJ, Michot F, Sielezneff I, Sastre B, Pigot F, Juguet F, Faucheron JL, Voirin D, Chipponi J. [Repair of rectocele using the Stapled TransAnal Rectal Resection (STARR) technique: intermediate results from a multicenter French study]. J Chir (Paris). 2008 Jan-Feb;145(1):27-31. doi: 10.1016/s0021-7697(08)70298-9. French. PMID 18438279
- [Background] Gagliardi G, Pescatori M, Altomare DF, Binda GA, Bottini C, Dodi G, Filingeri V, Milito G, Rinaldi M, Romano G, Spazzafumo L, Trompetto M; Italian Society of Colo-Rectal Surgery (SICCR). Results, outcome predictors, and complications after stapled transanal rectal resection for obstructed defecation. Dis Colon Rectum. 2008 Feb;51(2):186-95; discussion 195. doi: 10.1007/s10350-007-9096-0. Epub 2007 Dec 22. PMID 18157718
- [Background] Liu WC, Wan SL, Yaseen SM, Ren XH, Tian CP, Ding Z, Zheng KY, Wu YH, Jiang CQ, Qian Q. Transanal surgery for obstructed defecation syndrome: Literature review and a single-center experience. World J Gastroenterol. 2016 Sep 21;22(35):7983-98. doi: 10.3748/wjg.v22.i35.7983. PMID 27672293